CLINICAL TRIAL: NCT00407381
Title: Ranibizumab for Edema of the Macula in Diabetes: a Phase 2 Study ( The Read-2 Study)
Brief Title: The Ranibizumab for Edema of the mAcula in Diabetes-2 (READ-2) Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00005254
Record Dates: First submitted 2006-12-01; First posted 2006-12-05 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Diabetic Macular Edema
Keywords: DME
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ranibizumab (Experimental): Ranibizumab (RBZ) intravitreal injection alone
  Interventions: Drug: Ranibizumab
- Laser (Active Comparator): Laser photocoagulation
  Interventions: Procedure: Laser photocoagulation
- Laser with Ranibizumab (Experimental): Laser following intravitreal injection of RBZ
  Interventions: Drug: Ranibizumab; Procedure: Laser photocoagulation

INTERVENTIONS:
Drug: Ranibizumab — Ranibizumab for intravitreal injection. .05ml dosing at 30 day intervals and pro re nata (PRN) with dosing criteria.
  Other Names: Lucentis
  Arms: Laser with Ranibizumab; Ranibizumab
Procedure: Laser photocoagulation — Laser photocoagulation in either focal or grid pattern as determined by investigator.
  Arms: Laser; Laser with Ranibizumab

SUMMARY:
This study is being done to see if the investigational drug Ranibizumab (RBZ) given by injection into the eye, is safe and effective to use in people with diabetic macular edema (DME). The investigators want to compare RBZ to laser treatment which is the current standard way to treat DME.

RBZ blocks a growth factor that is thought to be involved in the formation of abnormal blood vessels that cause loss of vision in patients with DME.

DETAILED DESCRIPTION:
The READ-2 Study is a phase 2 randomized, multi-center clinical trial to be conducted under an investigator-initiated investigational new drug (IND). The study aims to enroll 126 patients, who will be randomized into 3 different groups. The primary objectives of the READ-2 Study are: (a) to obtain data on the bioactivity and dose interval effects of intravitreal ranibizumab (RBZ) alone, as well as in combination with laser photocoagulation, on retinal thickness and visual acuity in subjects with DME; and (b) to obtain additional safety and bioactivity data to aid in the design of a phase 3 clinical trial to evaluate ranibizumab as a therapeutic option for patients with DME The study consists of a 2-week screening period (Days -14 to 0), a 6-month treatment period with a primary time endpoint, and a 18-month follow-up and treatment period with secondary time endpoints. Consented subjects will enter the 14-day screening period to determine eligibility. Serum chemistry and hematology testing, urinalysis, pregnancy testing, and macular thickness measurements based on optical coherence tomography (OCT) will be performed. Screening will also include VA, ophthalmic examination and fluorescein angiography (FA) entry criteria.

Patients who have ETDRS visual acuity of 20/40 or worse, but better than or equal to 20/320 due to foveal thickening from macular edema secondary to diabetes (type 1 or 2) and who meet eligibility criteria will be eligible to enroll in the study. Baseline foveal thickness by OCT must be at least 250, which is often associated with VA of 20/40 or worse and which provides sufficient thickening so that a treatment effect is easily detectable (Nguyen et al. 2004). Approximately 126 patients with DME will be enrolled in this study from all clinical sites in the study. Every effort will be made to recruit and enroll eligible patients from men and women of all ethnic and social backgrounds. Patients who meet entry criteria will be able to enroll in the study until the quota of patients has been achieved.

ELIGIBILITY:
Inclusion:

* Signed informed consent and authorization of use and disclosure of protected health information
* Age greater than 18 years
* Diagnosis of diabetes mellitus (type 1 or type 2) and serum HbA1c greater than 5.5% within 12 months of randomization
* Retinal thickening secondary to diabetes mellitus (diabetic macular edema) involving the center of the fovea.
* Diagnosis must be confirmed by OCT images
* Foveal thickness of greater than 250, as assessed by OCT
* Best corrected visual acuity score in the study eye of 20/40 to 20/320 inclusive (Snellen equivalents using the ETDRS protocol at a distance of 4 meters). Only one eye will be treated in the study. If both eyes are eligible, the investigator will select the eye to be enrolled. Visual acuity in the non-study eye must be greater than 20/800.
* In the opinion of the investigator, decreased vision in the study eye is due to foveal thickening from DME and not from other obvious causes.
* In the opinion of the investigator, laser photocoagulation can be withheld for at least 30 days after the patient has enrolled in the study

Exclusion Criteria:

* Panretinal photocoagulation or macular photocoagulation within 3 months of study entry in the study eye
* Use of intraocular or periocular injection of steroids in the study eye (e.g., triamcinolone) within 3 months of study entry
* Previous participation in a study and receipt of anti-angiogenic drugs (pegaptanib sodium, ranibizumab, anecortave acetate, protein kinase C inhibitor, etc.) within 2 months of study entry
* Eyes in which the investigators do not feel appropriate to do any additional laser photocoagulation
* Proliferative diabetic retinopathy in the study eye, with the exceptions of inactive, fibrotic proliferative diabetic retinopathy that has regressed following pan-retinal laser photocoagulation or tufts of neovascularization elsewhere (NVE) less than one disc area with no vitreous hemorrhage
* Vitreomacular traction or epiretinal membrane in the study eye evident biomicroscopically or by OCT
* Structural damage to the center of the macula in the study eye likely to preclude improvement in visual acuity following the resolution of macular edema, including atrophy of the retinal pigment epithelium, subretinal fibrosis, laser scar(s), macular ischemia, or organized hard exudate plaque
* Ocular disorders in the study eye that may confound interpretation of study results, including retinal vascular occlusion, retinal detachment, macular hole, or choroidal neovascularization of any cause (e.g., age related macular degeneration (AMD), ocular histoplasmosis, or pathologic myopia)
* Concurrent disease in the study eye that could compromise visual acuity or require medical or surgical intervention during the first 6-month study period
* Eyes which are likely to need cataract surgery and intraocular lens implantation within the first 6 months of the study
* Cataract surgery in the study eye within 3 months of study entry; Yttrium-Aluminum-Garnet (YAG) laser capsulotomy within 2 months of study entry; or any other intraocular surgery within 3 months preceding Day 0.
* History of vitreoretinal surgery in the study eye within 3 months of study entry
* Uncontrolled glaucoma (defined as intraocular pressure greater than 30 mm Hg despite treatment with anti-glaucoma medications)
* Uncontrolled diabetes mellitus, as evidenced by glycosylated hemoglobin (HbA1c) value greater than 12%
* Premenopausal women not using adequate contraception
* Any women who are pregnant
* International normalized ratio (INR) greater than or equal to 3.0 (e.g. due to current treatment with warfarin). The use of aspirin or other anticoagulants is not an exclusion
* History of gastrointestinal bleeding within 2 months of study enrollment
* History of major gastrointestinal, cardiothoracic, gynecological, genitourinary, or orthopedic surgeries within 2 months of study enrollment
* History of cerebral vascular accident, myocardial infarction, transient ischemic attacks within 6 months of study enrollment
* Any patients who are on renal dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2006-12; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Do, MD, Principal Investigator — Truhlsen Eye Institute, University of Nebraska Medical Center
Locations (20):
- United States (20):
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - University of Southern California, Los Angeles, California
  - East Bay Retina Consultants, Oakland, California
  - Retina Institute of California, Pasadena, California
  - University of California, San Francisco, San Francisco, California
  - Yale Eye Center, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Illinois Retina Associates Rush University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - Wilmer Eye Institute at Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - New England Retina Consultants, PC, West Springfield, Massachusetts
  - Retinal Consultants of Nevada, Las Vegas, Nevada
  - University of New Mexico, Albuquerque, New Mexico
  - Duke Eye Center, Durham, North Carolina
  - Eye Care Specialists, PC, Kingston, Pennsylvania
  - Southern New England Retina Associates, Providence, Rhode Island
  - Black Hills Regional Eye Institute, Rapid City, South Dakota

REFERENCES:
- [Derived] Do DV, Nguyen QD, Khwaja AA, Channa R, Sepah YJ, Sophie R, Hafiz G, Campochiaro PA; READ-2 Study Group. Ranibizumab for edema of the macula in diabetes study: 3-year outcomes and the need for prolonged frequent treatment. JAMA Ophthalmol. 2013 Feb;131(2):139-45. doi: 10.1001/2013.jamaophthalmol.91. PMID 23544200

RESULTS

PARTICIPANT FLOW:
Groups:
- Ranibizumab Only: Ranibizumab (RBZ) intravitreal injection alone
  Ranibizumab: Ranibizumab for intravitreal injection. .05ml dosing at 30 day intervals and pro re nata (PRN) with dosing criteria.
- Laser Only: Laser photocoagulation
  Laser photocoagulation: Laser photocoagulation in either focal or grid pattern as determined by investigator.
- Laser With Ranibizumab (RBZ): Laser following intravitreal injection of RBZ
  Ranibizumab: Ranibizumab for intravitreal injection. .05ml dosing at 30 day intervals and PRN with dosing criteria.
  Laser photocoagulation: Laser photocoagulation in either focal or grid pattern as determined by investigator.
Period: Overall Study
Arm/Group | Ranibizumab Only | Laser Only | Laser With Ranibizumab (RBZ)
Started | 42 | 42 | 42
Completed | 39 | 38 | 40
Not Completed | 3 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Ranibizumab Only: RBZ intravitreal injection alone
  Ranibizumab: Ranibizumab for intravitreal injection. .05ml dosing at 30 day intervals and PRN with dosing criteria.
- Laser With RBZ: Laser following intravitreal injection of RBZ
  Ranibizumab: Ranibizumab for intravitreal injection. .05ml dosing at 30 day intervals and PRN with dosing criteria.
  Laser photocoagulation: Laser photocoagulation in either focal or grid pattern as determined by investigator.
- Total: Total of all reporting groups
Arm/Group | Ranibizumab Only | Laser Only | Laser With RBZ | Total
Number analyzed (Participants) | 42 | 42 | 42 | 126
Age, Continuous [Mean (Full Range); unit: years] | 62 [32 to 84] | 62 [34 to 86] | 62 [35 to 82] | 62 [32 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 23 | 22 | 74
  Male | 13 | 19 | 20 | 52

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA) at Month 6
Description: Mean change of best corrected visual acuity letters (BCVA) at month 6
Time Frame: 6 months
Population: Mean change in BCVA at month 6
Measure: Mean (Standard Deviation); unit: Mean letter change in BCVA
Groups:
- RBZ Alone: RBZ intravitreal injection alone
  Ranibizumab: Ranibizumab for intravitreal injection. .05ml dosing at 30 day intervals and PRN with dosing criteria.
- Laser Alone: Laser photocoagulation
  Laser photocoagulation: Laser photocoagulation in either focal or grid pattern as determined by investigator.
Arm/Group | RBZ Alone | Laser Alone | Laser With RBZ
Number analyzed (Participants) | 42 | 42 | 42
Mean letter change in BCVA | 7.24 (5.54) | -0.43 (4.56) | 3.8 (5.2)

ADVERSE EVENTS:
Time Frame: 6 Months
Groups:
- Laser With Ranibizumab: Laser following intravitreal injection of RBZ
  Ranibizumab: Ranibizumab for intravitreal injection. .05ml dosing at 30 day intervals and PRN with dosing criteria.
  Laser photocoagulation: Laser photocoagulation in either focal or grid pattern as determined by investigator.
Arm/Group | Ranibizumab Only | Laser Only | Laser With Ranibizumab
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 1/42
Other Adverse Events (participants affected / at risk) | 1/42 | 4/42 | 3/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranibizumab Only (N=42) | Laser Only (N=42) | Laser With Ranibizumab (N=42)
Cerebrovascular Event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranibizumab Only (N=42) | Laser Only (N=42) | Laser With Ranibizumab (N=42)
Vitreous Hemorrhages (Eye disorders) | 1 (1) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No